CLINICAL TRIAL: NCT06322485
Title: An Online Self-management Intervention for Patients With Hand Fibromyalgia - a Randomized Controlled Trial
Brief Title: Online Self-management in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University (Other)
Collaborators: Fibrocentrum (Unknown)
Responsible Party: Principal Investigator, Andrea W.M Evers, PhD, Professor, Leiden University
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P16.230
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Fibromyalgia
Keywords: internet-based cognitive-behavioral therapy; cognitive-behavioral therapy; web-based; self-management; fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Masking Description: Blinding of participants and practitioners is not possible due to the nature of the study. However, the statistician who creates the randomization schedule and performs statistical analyses is blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based self-management intervention (Experimental): At the beginning of the treatment, a face-to-face introductory meeting is scheduled between the participant and a psychologist, where treatment goals will be set. Afterwards, a tailored self-management intervention, based on cognitive-behavioral methods, will be offered via an internet-based program. The psychologists offering the treatment have been trained in the tailored cognitive-behavioral protocol. One month and 2,5 months after finishing the online program, patients will be contacted by their treating psychologist for two booster sessions via telephone. Patients' goals will be evaluated and strategies to strengthen the achieved results will be discussed.
  Interventions: Behavioral: Internet-based self-management intervention
- Waitlist (No Intervention): Patients in the control condition will be assigned to a waiting list and will receive the internet-based self-management intervention after the active treatment group (after 6 months).

INTERVENTIONS:
Behavioral: Internet-based self-management intervention — An internet-based cognitive-behavioral therapy with six modules.
  Arms: Internet-based self-management intervention

SUMMARY:
This study has been previously registered with the National Trial Registry (NTR6267) that has been cancelled. The registered trial has been automatically transferred to a new "Landelijk Trial Register", which does not contain all correct information on the current study and where no corrections can be made. Hence, the current study has been registered again with ClinicalTrials.gov.

The goal of this clinical trial is to study the effectiveness of an internet-based self-management intervention in adult patients with fibromyalgia. A randomized controlled trial (RCT) will be performed, in which 70 participants will be randomized to either the self-management intervention or a waitlist control condition (patients in the waitlist condition will receive the intervention after the intervention ends in the intervention group, i.e., after 6 months). The primary effect constitutes of the difference in change in pain coping between patients in the intervention and control condition from baseline to post-intervention. As secondary outcomes, a number of other psychological and physical outcome measures will be assessed (e.g., health-related quality of life, well-being, pain impact on daily life, pain cognitions). Also, cost-effectiveness of the intervention and the quality of the therapeutic relationship will be measured.

DETAILED DESCRIPTION:
Rationale: Fibromyalgia has a high clinical burden, with patients experiencing considerable pain, physical disability, and an often decreased health-related quality of life (HR-QoL). Improving patients' skills in managing a chronic condition ("self-management") is increasingly recognized as vital in the treatment of somatic conditions and is becoming more common in clinical practice and research. In this study, the effectiveness of an internet-based self-management intervention focusing on coping skills related to chronic pain compared with a waitlist control condition is studied.

Objective: To study the effectiveness of the internet-based self-management intervention in patients with fibromyalgia.

Study design: An RCT will be performed, in which 70 patients will be randomized to either the internet-based self-management intervention or a waitlist control group. Baseline, post-intervention, 6-week, and three-month follow-up questionnaires will be used to measure primary and secondary outcomes.

Study population: Patients ≥18 years diagnosed with fibromyalgia (confirmed by their general practitioner or a medical specialist) who visit the 'Fibrocentrum', a fibromyalgia treatment centre in Leiden, The Netherlands, will be invited to participate in the study. Patients need to have a pain duration of a minimum of 3 months, be fluent in Dutch, be able to give informed consent, and own a computer with internet access. Difficulties with (written) communication and internet literacy, severe physical and psychiatric comorbidities that interfere with the study protocol (e.g., addiction, psychosis, and suicidal ideation), pregnancy, on-going psychological treatment elsewhere, and participation in other clinical trials are exclusion criteria.

Intervention: The cognitive-behavioral intervention begins with a face-to-face intake session in which personal goals for the intervention are set. Afterwards, the tailored self-management intervention, consisting of 6 modules, will be offered via an internet-based program. The first introductory module includes goal-setting and the last module includes relapse prevention; the four modules in between focus on learning how to cope with the consequences of a chronic condition in daily life. The topics of the modules are (1) activity, (2) mood, (3) thoughts, and (4) the social environment. At least once a week, a psychologist provides participants with feedback and motivational support through messages in a secured mail box in the internet-based program. After finishing the internet-based intervention, two booster sessions will take place via telephone (1 month and 2,5 months after the program). Patients will be called by their psychologist and their goals will be evaluated and strategies to strengthen the achieved results will be discussed.

Main study parameters/endpoints: The primary effect will be determined by comparing the VAS pain coping scores after the intervention between the waitlist control group and intervention group, corrected for baseline VAS pain coping scores. As secondary outcomes, several other psychological and physical outcomes will be measured (e.g., HR-QoL, pain cognitions, pain impact on daily life, well-being), as well as quality of the therapeutic relationship and cost-effectiveness of the intervention.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In the waitlist control condition, patients will receive the intervention after the intervention ends in the intervention group (after 6 months). In the intervention group patients will be offered an internet-based self-management intervention, which could improve their pain coping and other psychological and physical outcomes. No risk is involved with participation in this study. The only burden for participants is time investment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with fibromyalgia, as previously confirmed by their treating general practitioner or a medical specialist.
2. Pain complaints with a minimal duration of 3 months.
3. Minimum age of 18 years.
4. Fluent in Dutch.
5. Able to give informed consent.
6. Own a computer with internet access.

Exclusion criteria:

1. Difficulties with (written) communication (e.g., due to analphabetism) and with internet literacy.
2. Severe physical and psychiatric comorbidities that interfere with the study protocol, such as psychosis, addiction, suicidal ideation.
3. On-going psychological treatment elsewhere.
4. Participation in other clinical trials.
5. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Change in pain coping | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  A visual analogue scale (VAS) from 0 to 10 will be used to measure pain coping, with higher scores indicating better pain coping. The primary endpoint is the difference in change in pain coping between patients in the intervention and control condition from baseline to post-intervention (immediately after the intervention).

SECONDARY OUTCOMES:
Change in well-being | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  A VAS from 0 to 10 will be used to measure well-being, with higher scores indicating better well-being.
Change in illness cognitions | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  Illness cognitions will be assessed by the Illness Cognition Questionnaire (ICQ; using Helplessness and Acceptance scales). Items are scored on a 4-point Likert scale ranging from "not at all" to "completely". Higher scale scores reflect greater use of the assessed construct.
Change in pain coping strategies | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  Pain coping strategies will be assessed by the Pain Coping Inventory (PCI) that comprises six scales, namely, Pain Transformation, Distraction, and Reducing Demands (three active pain coping strategies), and Retreating, Worrying, and Resting (three passive pain coping strategies). Items are scored on a 4-point Likert scale ranging from "hardly ever" to "very often". Higher scale scores reflect greater use of the assessed pain coping strategy.
Change in Illness Perceptions | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  Illness perceptions will be assessed by the Illness Perception Questionnaire (IPQ-R). The Identity scale consists of the sum of yes-rated items (patients rate whether they believe certain symptoms to be related to their illness). Furthermore, the remaining scales described below are rated on a 5-point Likert type scale ranging from "strongly disagree" to "strongly agree". High scores on the Timeline Acute/Chronic and Cyclical, Consequences, and Emotional Representations scales indicate beliefs about the chronicity and cyclical nature of the illness, the negative consequences of the illness, and patients' emotional experience of their illness. High scores on the Personal and Treatment Control and Illness Coherence scales reflect positive beliefs about perceived control and an understanding of the illness.
Change in pain | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  A VAS ranging from 0 to 10 will be used to measure pain, with higher scores reflecting more severe pain.
Change in pain interference in daily functioning and pain severity, and as exploratory measures support, life control, and affective distress | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  Part 1 of the Multidimensional Pain Inventory-Dutch Language Version (MPI-DLV) will be used with Interference and Pain Severity scales and as exploratory measures Support, Life Control, and Affective Distress. Items are rated on different 7-point Likert scales, with higher scores reflecting greater intensity in a subscale.
Change in health-related quality of life | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  Health-related quality of life will be assessed with the RAND-36, which consists of 36 items that are averaged, resulting in eight health scale scores, namely Physical Functioning, Role Limitations due to Physical Health Problems, Role Limitations due to Personal or Emotional Problems, Social Functioning, Emotional Well-being, Energy/Fatigue, Bodily Pain, and General Health Perceptions. The questionnaire also includes one item on perceived change in health. Besides, physical and mental health composite scores will be calculated. Higher scores reflect more favorable health states.
Change in fibromyalgia impact | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  The Fibromyalgia Impact Questionnaire (FIQ) consists of 10 self-rated items covering the impact of fibromyalgia on different aspects of functioning and well-being. Total scores range from 0 to 100, with higher scores reflecting worse fibromyalgia impact.
Change in health-related quality of life | Baseline, immediately after the intervention, at 3 months follow-up.
  Health-related quality of life will be assessed by the Five-Level Version of the EQ-5D (EQ-5D-5L). In this questionnaire, 5 dimensions are measured in 5 items: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. A 5-point Likert scale ranging from "no problems" to "extreme problems" is used for every dimension, with higher scores reflecting more problems in a dimension. A VAS ranging from 0 to 100 (0 = "The best health you can imagine" to 100 = "The worst health you can imagine") is applied as well, with higher scores indicating a better health state as perceived by the patient.

OTHER OUTCOMES:
Economic evaluation: Five-Level Version of the EQ-5D (EQ-5D-5L) | Baseline, immediately after the intervention, at 3 months follow-up.
  The intervention will be economically evaluated with the Five-Level Version of the EQ-5D (EQ-5D-5L). Five items cover 5 dimensions of health-related quality of life: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. A 5-point Likert scale ranging from "no problems" to "extreme problems" is used in the questionnaire, with higher scores indicating more issues in a dimension. The 5 dimensions can be summed into a health state and utility values can be calculated for these health states.
Economic evaluation: iMTA Medical Consumption Questionnaire (iMCQ) | Baseline, immediately after the intervention, at 3 months follow-up.
  The intervention will be economically evaluated with the iMTA Medical Consumption Questionnaire (iMCQ), which measures health-care utilization.
Economic evaluation: iMTA Productivity Cost Questionnaire (iPCQ) | Baseline, immediately after the intervention, at 3 months follow-up.
  The intervention will be economically evaluated with the iMTA Productivity Cost Questionnaire (iPCQ). Productivity losses are assessed in three modules in this questionnaire, so that certain types of productivity losses can be omitted when these are not applicable to a population.
Patient satisfaction | Immediately after the intervention.
  The experience and satisfaction of patients with the intervention, and the perceived effect of the intervention will be assessed with an evaluation questionnaire comprising various numerical rating scales, Likert scales, and open questions.
Expected/perceived patient-provider interaction | Baseline and immediately after the intervention.
  The Internet-specific Therapeutic Relationship Questionnaire (ITRQ) will be used to assess the expected/perceived patient-provider interaction. The ITRQ comprises 10 items that are measured on a 10-point Likert scale ranging from "totally disagree" to "completely agree". The questionnaire consists of two scales (Internet-specific Time and Attention and Internet-specific Reflection and Comfort) and a total score. Higher scores reflect a stronger therapeutic relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Evers, PhD, Principal Investigator — Leiden University
Locations (1):
- Fibrocentrum, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Once an article on the study is published, a publication package will be published on DataverseNL. This package includes the manuscript, procedures, raw data files, computer code, and processed data files.
Supporting Information: SAP
Time Frame: Individual participant data (IPD) will become available once an article on the study is published on DataverseNL; the statistical analysis plan will be published on ClinicalTrials.gov during registration (the plan was developed before data analysis takes place).
Access Criteria: Open access.

REFERENCES:
- [Derived] Terpstra JA, van Beugen S, van der Vaart R, van Eersel RA, Dusseldorp E, Kloppenburg M, Evers AWM. An internet-based cognitive-behavioral self-management intervention for patients with hand osteoarthritis or fibromyalgia - Two randomized controlled trials. Internet Interv. 2026 Jan 19;43:100908. doi: 10.1016/j.invent.2026.100908. eCollection 2026 Mar. PMID 41631249

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT06322485/SAP_000.pdf